CLINICAL TRIAL: NCT01045213
Title: Phase 3 Study of the Efficacy of Proactive Integrated Care in Advanced COPD Patients Located in Areas With High COPD-related Mortality
Brief Title: Integrated Care Program for Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-0588; 09 FLA 000317 (Other: CHPHE)
Record Dates: First submitted 2010-01-06; First posted 2010-01-08 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Delivery of Health Care, Integrated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Proactive Integrated Care (Experimental): COPD education, self-management education, remote monitoring (Health Buddy, pulse oximeter, pedometer, spirometer) and enhance communication with cell phone contact with a coordinator.
  Interventions: Other: Integrated Care

INTERVENTIONS:
Other: Integrated Care — Study looking at the efficacy of a combination of Guideline-based COPD education, self-management training, remote telemonitoring and enhanced communication with a coordinator.

SUMMARY:
Integrated eHealth is an innovative, proactive approach to the management of patients with chronic cardiopulmonary disease. Our overall goal is to improve the health of patients by integrating guideline-based education, remote disease monitoring, coordinator-based disease management and healthcare provider-initiated therapy. Patients enrolled in the program receive a set of equipment, including a Health Buddy® telemonitor that connects to a normal telephone, as well as instruments to measure oxygen levels (pulse oximeter), lung function (spirometer) and activity (pedometer). Through the Health Buddy® patients receive guideline-based disease education in their own homes. The Health Buddy® also allows patients to transmit daily information about their symptoms, oxygen levels, lung function and ability to walk to program coordinators located at the University of Colorado Hospital. Our program coordinators are highly experienced nurses or respiratory therapists with expertise in the management of chronic obstructive pulmonary disease (COPD) and congestive heart failure (CHF). Through this remote disease education/monitoring program, patients learn to take a more active role in the management of their own disease. However, once the coordinators identify early warning signs of a potential problem, patients are contacted and connected to their primary healthcare provider for early intervention. By this integrated approach to care, patients learn self-management techniques, physician communication is enhanced, and early interventions for problems are possible. We propose to target the Integrated eHealth Program to areas of Colorado that are highly impacted by COPD.

Key Objectives: The key objectives are to improve COPD care in the 16 Colorado counties with high COPD mortality rates.

Target Population: We will target patients with severe or very severe COPD.

Expected Outcomes: We expect that this study will increase the use of evidence-based guidelines in the screening, diagnosis and treatment of COPD, resulting in improved quality-of-life and a reduction in healthcare utilization.

ELIGIBILITY:
Inclusion Criteria:

* COPD Diagnosis by Gold Guidelines
* Airflow obstruction on spirometry defined by an FEV1/FVC less than or equal to 70% and an FEV1 less than 50% predicted, or and FEV1 greater than or equal to 50% predicted with a history of a COPD exacerbation within one year, or an FEV1 greater than or equal to 50% predicted and on long-term oxygen therapy.
* Standard land-line telephone
* Legal US residency status residing in Adams, Alamosa, Bent, Crowley, Dolores, El Paso, Fremont, Kiowa, Logan, Morgan, Montezuma, Otero, Prowers, Rio Blanco, or Washington counties in Colorado

Exclusion Criteria:

* Asthma
* Co-existing conditions that are likely to cause death within two years. Patients with CXR evidence of interstitial lung disease, or other pulmonary diagnoses at the time of enrollment, aside from COPD-related bronchiectasis. Patients with end-stage liver, renal or muscle disease, HIV, or a diagnosis of dementia.
* Participation in another treatment study
* Inability or unwillingness to cooperate with self-monitoring and reporting components
* Prisoners, pregnant women, institutionalized patients
* Current alcohol or drug abuse
* Non-English speakers
* Inability to complete a consent
* Illegal alien, non-Colorado resident, or non-resident of targeted counties

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Quality of Life measured by the St. Georges Respiratory Questionnaire | 3 months

SECONDARY OUTCOMES:
Guideline-based medical care | 3 months
Oxygen utilization and pre/post exercise oxygen saturations | 3 months
Smoking status | 3 months
Exercise status measured by the 6 minute walk test | 3 months
Symptoms including cough, sputum production and dyspnea (measured by the modified Medical Research Council (MMRC) dyspnea scale) | 3 months
Body Mass Index, Obstruction, Dyspnoea, Exercise Capacity (BODE) Index | 3 months
Healthcare utilization | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: William Vandivier, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States